CLINICAL TRIAL: NCT07387718
Title: Artificially Intelligent Robot (AIR) Support for Pediatric Asthma Education
Brief Title: AIR Support: Artificially Intelligent Robot (AIR) Support for Pediatric Asthma Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Cynthia Foronda, Assistant Dean for Innovation and Clinical Scholarship, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20251352
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Asthma in Children; Artificial Intelligence
MeSH Terms: interventions — Air

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Asthma Education (Control) (Active Comparator): Participants in this arm will receive one standard asthma education session during a single clinic visit lasting approximately 5 minutes.
  Interventions: Behavioral: Standard Asthma Education
- Standard Education Plus Artificially Intelligent Robot (AIR) Support Intervention (Experimental) (Experimental): Participants in this arm will receive standard asthma education plus one artificially intelligent robot supported education session during a single clinic visit lasting approximately 15 minutes.
  Interventions: Behavioral: Standard Asthma Education; Behavioral: Artificially Intelligent Robot (AIR) Support Intervention

INTERVENTIONS:
Behavioral: Standard Asthma Education — Participants will receive the usual asthma education provided by their healthcare provider during the clinic visit, including asthma action plan and metered dose inhaler and spacer teaching..
Behavioral: Artificially Intelligent Robot (AIR) Support Intervention — Participants will receive a single 15-minute robotic asthma education session delivered by the Artificially Intelligent Robot/Human Support Robot (AIR/HSR).
  Arms: Standard Education Plus Artificially Intelligent Robot (AIR) Support Intervention (Experimental)

SUMMARY:
The purpose of this prevention study is to evaluate the design and usability of a newly developed asthma education protocol with the Human Support Robot (HSR) for children with asthma.

ELIGIBILITY:
Inclusion (Eligibility) Criteria for Caregivers or Parents:

* The participant must be at least 18 years old.
* The participant must be willing and able to participate.
* The participant can read English or Spanish and is able to fill out survey instruments by themselves or with assistance.
* The participant cares for a child with asthma.

Exclusion (Eligibility) Criteria for Caregivers or Parents:

* The participant is younger than 18 years old.
* The participant is unwilling to participate in the study.
* The participant is unable to complete survey instruments.
* The participant does not care for a child with asthma.

Inclusion (Eligibility) Criteria for Children:

* The participant must be at least 3 years old - 17 years old with asthma.
* The participant must assent to participation.
* The participant's guardian must have consented.

Exclusion (Eligibility) Criteria for Children:

* The participant is younger than 3 years old.
* The participant does not have asthma.
* The participant is unwilling to participate in the study.
* The participant's guardian did not consent.

Inclusion (Eligibility) Criteria for Healthcare Providers:

* The participant must be at least 18 years old.
* The participant must be willing and able to participate.
* The participant can read English and is able to fill out survey instruments by themselves.
* The participant must view a robotic education session.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Human Support Robot: Enrollment Rate | Immediately after robotic session and up to 3 months afterwards via recordings and documentation.
  Feasibility will be assessed by measuring the enrollment rate for the study involving the Human Support Robot. Enrollment rate will be calculated as the number of participants enrolled divided by the number of eligible participants approached, expressed as a percentage. Higher percentages indicate greater feasibility of implementation.
Feasibility of the Human Support Robot: Completion Rate | Immediately after robotic session and up to 3 months afterwards via recordings and documentation.
  Feasibility will be evaluated by measuring the completion rate for the study procedures involving the Human Support Robot. Completion rate will be calculated as the number of enrolled participants who complete all required study procedures - including the education session, survey, inhaler-use demonstration, and interview - divided by the total number of participants enrolled, expressed as a percentage. Higher percentages indicate greater feasibility of implementation.
Feasibility of the Human Support Robot: Session Length | Immediately after robotic session and up to 3 months afterwards via recordings and documentation.
  Feasibility will be measured by recording the duration in minutes of the robot education session. More consistent and shorter session durations indicate better feasibility for clinic workflow and integration of the Human Support Robot.
Feasibility of the Human Support Robot: Number of Technical Issues | Immediately after robotic session and up to 3 months afterwards via recordings and documentation.
  Feasibility will be assessed by recording the number and type of technical issues occurring during the robot-supported education session, including hardware malfunctions, software errors, or disruptions requiring staff assistance. Fewer technical issues indicate greater feasibility of implementing the Human Support Robot in a clinic setting.
Acceptability of the Human Support Robot or Acceptability of the Robot-Supported Education Session | Immediately after the robotic session (same clinic visit) and up to 3 months afterwards via recordings and documentation.
  Acceptability of the robot will be evaluated by using the Technology Acceptance Model Questionnaire. The questionnaire includes items assessing perceived usefulness and perceived ease of use, each rated on a 7-point Likert scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"). Scores will be averaged to produce subscale scores ranging from 1 to 7, with higher scores indicating greater acceptability.

SECONDARY OUTCOMES:
Child Engagement (PROMIS) | Day 1
  Child engagement will be evaluated using a slightly adapted Patient-Reported Outcomes Measurement Information System (PROMIS) Early Childhood Parent Engagement measure. This questionnaire includes items assessing the child's attention, interest, and participation during activities. Each item is rated on a 5-point Likert scale ranging from 1 ("never") to 5 ("always"). Item responses are summed and converted to a standardized T-score (mean = 50, standard deviation = 10). Higher T-scores indicate greater engagement.
Child inhaler technique (Coaching Tool) | Day 1
  Child knowledge will be assessed using the Inhaler Technique Coaching Tool, a structured checklist evaluating each step of proper inhaler use. The research assistant will score each step as correct (1) or missed or done improperly (0). Scores will be summed to produce a total score ranging from 0 - 6, with higher scores indicating more accurate inhaler technique and greater knowledge of inhaler use.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Foronda, PhD, Principal Investigator — University of Miami
Locations (1):
- Batchelor Children's Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pasternak K, Foronda C, Downs C, Visser U. Social robots for pediatric asthma education: A pilot study. In: Staffa M, et al., eds. Social Robotics + AI. ICSR+AI 2025. Lecture Notes in Computer Science. Vol 16131. Singapore: Springer; 2026. doi:10.1007/978-981-95-2379-5_35
- [Background] Foronda CL, Susas T, Castaño Cubillos N, Pasternak K, Downs CA, Visser U. Preparing nurses for the technological future: Robotic integration in nursing education. Teaching and Learning in Nursing. 2025. doi:10.1016/j.teln.2025.11.034
- [Background] Foronda C, Gonzalez JM, Snowden K, Prather S, Majilton C, Weisman A, Parmeter S, Herrera A, Gattamorta KA, Gonzalez JE, Downs C, Hooshmand M, Cardenas M. Improving knowledge and decreasing depressive symptoms in caregivers of children with asthma through the asthma academy: A randomized controlled trial. Int J Nurs Stud Adv. 2021 Oct 9;3:100047. doi: 10.1016/j.ijnsa.2021.100047. eCollection 2021 Nov. PMID 38746721